CLINICAL TRIAL: NCT01387880
Title: Phase II Examination of Irinotecan, Cetuximab and Everolimus to Chemotherapy Resistent Patients With Metastatic Colorectal Cancer and KRAS Mutations or After Progression With KRAS Wildtype on Irinotecan and Cetuximab - Effect and Biological Markers
Brief Title: Irinotecan, Cetuximab and Everolimus to Patients With Metastatic Colorectal Cancer
Acronym: ICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Benny Vittrup Jensen, onsultant, Herlev Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI 0923 ICE
Record Dates: First submitted 2011-06-27; First posted 2011-07-06 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Third line therapy; Fourth line therapy; KRAS mutation status; Cetuximab; Everolimus; Irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab, everolimus, irinotecan (Experimental)
  Interventions: Drug: Everolimus
- Cetuximab, everolimus and Irinotecan. (Active Comparator): Patients with metastatic colorectal cancer with KRAS mutant tumours are treated with cetuximab, everolimus and irinotecan.
  Patients with KRAS wildtype colorectal cancer that have progressed on therapy with cetuximab and irinotecan are treated with cetuximab, irinotecan and everolimus.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Patients with KRAS mutant tumours are treated with cetuximab, everolimus and irinotecan as third line.
  Patients with KRAS wildtype tumours that have progressed on therapy with cetuximab and irinotecan are treated with cetuximab, everolimus and Irinotecan.
  Arms: Cetuximab, everolimus, irinotecan
Drug: Everolimus — 1.66 mg per day up to 7½ mg per day

SUMMARY:
This is an open, multicenter phase II trial of therapy with a combination of cetuximab, and irinotecan every second week combined with a daily dose of everolimus to patients with metastatic colorectal cancer with Kirsten rat sarcoma viral oncogene (KRAS) mutation or to patients resistent to cetuximab and irinotecan therapy for metastatic colorectal cancer.

DETAILED DESCRIPTION:
Main objective:

* Number of patients with progressive disease that obtain disease control defined as the sum of patients that obtain a Complete Remission (CR), Partial Remission(PR, or stable disease (SD))

Secondary objectives:

* Time to progression after first therapy.
* Length of disease control (CR, PR and SD)
* Survival from date of start of therapy.
* Safety and toxicity of the therapy graded according to Common Toxicity Criteria version 3.0
* Influence of smoking on disease control, response, survival and time to progression and other effect parameters in the investigation.
* Significance of metabolic response evaluated by a Photon Emissions Tomography (PET)/Computer Tomography(CT)scan.
* Blood: Examine the influence of potential predictive and prognostic tumour biomarkers in blood as lactate dehydrogenase (LDH), Carcinoembryonic antigen (CEA), Vascular endothelial growth factor (VEGF), epidermal growth factor receptor (EGFR), Human Epidermal growth factor Receptor 2 (HER-2), YKL-40, Interleukin-6 (IL-6) ,metallopeptidase inhibitor 1 (TIMP-1), procollagen type I N-terminal propeptide (PINP), Procollagen type 3 N-terminal propeptide (P3NP), gen-, micro-ribonucleinate (microRNA)- and protein array profiles, metabolomics and C-reactive protein (CRP) 2 weeks after start of therapy and thereafter every 8.weeks on disease control, response, survival and time to progression and other parameters investigated.
* Tissue: Examine possible predictive and prognostic biomarkers in tissue from primary tumour or metastases for micro-RNAarray profiles, mutations in K-RAS, murine sarcoma viral oncogene homolog (BRAF), Phosphoinositide 3-kinase (PIK3CA), EGFR, tumor protein 53 (p53), and protein expression and polymorphisms of th phosphatase and tensin homolog (PTEN), epiregulin (EREG), amphiregulin (AREG), Insulin-like growth factor 1 (IGF-1), IGF-1 Receptor (IGF-1R), VEGF, p53, topoisomerase 1 (Topo1), YKL-40, and TIMP-1
* Correlation between possible predictive and prognostic biomarkers in blood and tissue.

ELIGIBILITY:
Criteria for inclusion:

* Patients with a histological or cytological verified adenocarcinoma of the colon or rectum with non-resectable or metastatic cancer.
* Patients with measurable disease without previous radiotherapy
* Patients with metastatic colorectal cancer with progression after previous therapy with 5-fluoropyrimidines, oxaliplatin or irinotecan. Patients should have been treated with oxaliplatin, but if oxaliplatin has be contraindicated or not tolerated the patient can participate in the trial.
* Patients with KRAS-mutation in their primary tumour or metastasis.
* Patients with progression after therapy with irinotecan or cetuximab independent of KRAS mutation status.
* Previous radiotherapy is allowed to less than 25 % of the bone marrow.
* Age more or equal to 18 years.
* Performance status less than 3.
* An expected survival time of at least 3 months.
* Signed informed consent according to specifications from the ethical comites.

Criteria for exclusion:

* Former or other concurrent malignant disease except treated basal cell carcinoma or in situ cervical cancer.
* No cytotoxic therapy or other experimental treatment within 28 days before inclusion.
* No former therapy with everolimus or other rapamycin as sirolimus or temsirolimus.
* No known hypersensitivity for one or more components in the therapy.
* No uncontrolled diabetes
* No serious non-healing wounds, gastric ulcers, bone fractures, greater surgical procedures, major traumatic injuries within 28 days before inclusion.
* No ongoing bleeding or pathological condition associated with a risk of bleeding.
* No liver disease as cirrhose, chronical active hepatitis or chronic persistent hepatitis.
* No gastrointestinal disturbances in function that might cause a major change in the absorption of everolimus as ulcerative disease, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome.
* No planned immunisation with attenuated virus in the study period.
* Patients that is unable to follow treatment or evaluation plan.
* Every condition or therapy that after the judgement of investigator might infer the patient a risk or influence the trials objective.
* Pregnant or breastfeeding women.
* At fertile women this is insured by a negative test of pregnancy or use of a safe anticonception during the trial period and at least 3 months after end of treatment.
* Patients with active infections or other serious medical co-morbidity, that might prevent the patient from being treated with the protocoled therapy.
* Incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Clinical benefit (SD+PR+CR) | 1 year
  Clinical benefit is defined as the number of patients with stable disease lasting 2 months and partial response and CR as defined in RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Benny V Jensen, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Herlev University Hospital, Herlev, Copenhagen, Denmark

REFERENCES:
- [Derived] Spindler KG, Demuth C, Sorensen BS, Johansen JS, Nielsen D, Pallisgaard N, Hoegdall E, Pfeiffer P, Vittrup Jensen B. Total cell-free DNA, carcinoembryonic antigen, and C-reactive protein for assessment of prognosis in patients with metastatic colorectal cancer. Tumour Biol. 2018 Nov;40(11):1010428318811207. doi: 10.1177/1010428318811207. PMID 30486767